CLINICAL TRIAL: NCT03162120
Title: A Single Site, Interventional, Comparative Study to Evaluate the Safety and Efficacy of Ranolazine Plus Metoprolol Combination vs. FlecainidE pluS Metoprolol Combination in ATrial Fibrillation Recurrences
Brief Title: Comparison of Effectiveness of Ranolazine Plus Metoprolol Combination vs. FlecainidE pluS Metoprolol Combination in ATrial Fibrillation Recurrences FOllowing PhaRmacological or Electrical CardioverSion of AtRial Fibrillation
Acronym: PRESERVE-SR
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: new study type, it will be re-organiZed as an Investigator Initiated Study (IIS)
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIS-EL-VASS-2017
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation; Recurrence
MeSH Terms: conditions — Atrial Fibrillation; Recurrence | interventions — Ranolazine; Flecainide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranolazine plus Metoprolol Combination (Active Comparator): Ranolazine plus Metoprolol Combination in ATrial Fibrillation Recurrences FOllowing PhaRmacological or Electrical CardioverSion of AtRial Fibrillation
  Interventions: Drug: Ranolazine plus Metoprolol Combination
- FlecainidE pluS Metoprolol Combination (Active Comparator): FlecainidE pluS Metoprolol Combination in in ATrial Fibrillation Recurrences FOllowing PhaRmacological or Electrical CardioverSion of AtRial Fibrillation
  Interventions: Drug: FlecainidE pluS Metoprolol Combination

INTERVENTIONS:
Drug: Ranolazine plus Metoprolol Combination — Ranolazine plus Metoprolol Combination in ATrial Fibrillation Recurrences FOllowing PhaRmacological or Electrical CardioverSion of AtRial Fibrillation
  Other Names: RM group
  Arms: Ranolazine plus Metoprolol Combination
Drug: FlecainidE pluS Metoprolol Combination — FlecainidE pluS Metoprolol Combination in ATrial Fibrillation Recurrences FOllowing PhaRmacological or Electrical CardioverSion of AtRial Fibrillation
  Other Names: FM group
  Arms: FlecainidE pluS Metoprolol Combination

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia in clinical practice with a prevalence reaching 5% in patients older than 65 years and an incidence that increases progressively with age.1 According to the most recent guidelines, class Ic anti-arrhythmic drugs are considered the first line treatment in patients without significant structural heart disease. Flecainide is effective in preventing AF recurrences in 31-61% of cases according to different studies.2-5 A recent study showed that the combination of Flecainide and Metoprolol improves effective rhythm control in patients with persistent symptomatic AF compared to Flecainide or Metoprolol alone.6 In contrast, the combination of Flecainide and Metoprolol conferred no significant benefit over Flecainide alone in patients with paroxysmal AF. This suggests different underlying mechanisms for paroxysmal and persistent AF. Pulmonary veins are likely the main focus triggering paroxysmal AF while in persistent AF the role of pulmonary veins is less important.

DETAILED DESCRIPTION:
Ranolazine (RN) is a novel antianginal agent with increasingly appreciated antiarrhythmic properties that can suppress ventricular and supraventricular arrhythmias including AF. The antiarrhythmic actions of RN are mainly attributed to its ability to block INa, INaL, and the rapidly activating delayed rectifier potassium current (IKr).7 In experimental studies, RN proved very effective in suppressing late phase 3 early afterdepolarization and delayed afterdepolarization mediated triggered activity in pulmonary vein sleeves.8 RN was shown very effective in suppressing persistent, vagally mediated AF in animal models.9 Clinical evidence of an AF-suppressing effect of RN comes mainly from small caliber studies. Murdock et al, reported a high conversion rate (72%) after administration of 2,000 mg of RN (in a "pill-in-the-pocket" fashion) in patients with short lasting (<48 hours) new onset paroxysmal AF.10 Our group demonstrated both the superior efficacy and the accelerated action of the combined therapy of Amiodarone with RN compared to Amiodarone alone in patients with paroxysmal AF. Notably, the efficacy benefit of this combination was more pronounced in patients with dilated left atria which is also more likely to occur in cases of persistent AF.11, 12 In a prospective, randomized, double-blind, placebo-control phase II study, different doses of RN were tested in the prevention of AF recurrence after successful electrical cardioversion. Despite the fact that the study did not reach its primary end-point since none of the individual doses of RN significantly delayed the time to first AF recurrence as compared with placebo, an antiarrhythmic efficacy for the two higher doses of RN (500 and 750mg bd) was strongly suggested. The same study confirmed the safety of RN with no evidence for proarrhythmia.13 Notably, beta-blockers were used in less than 50% of patients studied in this study.

Although the efficacy of beta-blockers in the maintenance of sinus rhythm is low, the addition of a beta-blocker to an antiarrhythmic agent that exerts its action by inhibiting inward Na+ current like RN and Flecainide may represent an interesting approach in preventing AF relapse. Various laboratory studies have demonstrated that inward Na+ current could be modulated by beta-adrenergic receptors in a variety of cell lines.14, 15 In this context, the beta-blocking activity of Amiodarone or Dronedarone may account for the successful combination with RN in suppressing AF in either experimental or clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* patients with AF
* recently converted to sinus rhythm (>24hrs and < 7 days)
* admitted in the 3rd University Cardiology Clinic of Ippokrateion Hospital
* eligible to participate in the study and follow the study procedures
* signed informed consent

Exclusion Criteria:

* use of IC antiarrhythmic agents or
* Sotalol during the last 48 hours,
* chronic use of oral or intravenous Amiodarone for the last 48 hours,
* recent acute coronary syndrome,
* heart failure New York Heart Association class III or IV,
* severe left ventricular dysfunction with left ventricular ejection fraction <40%,
* atrioventricular conduction disorders (atrioventricular block,
* complete left bundle branch block and bi-fascicular block),
* heart rate < 50 bpm,
* sick sinus syndrome,
* thyroid dysfunction and severe pulmonary, renal, or
* liver disease
* - not eligible to participate in the study and follow the study procedures
* no signed informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of 1-year-recurrences | 12 months
  efficacy and safety of the combination of RN and Metoprolol vs. the combination of Flecainide and Metoprolol in preventing AF recurrences during a 1-year follow-up period in patients with AF of longer than 24-hour duration who were cardioverted to sinus rhythm either pharmacologically or electrically

SECONDARY OUTCOMES:
Number of 48-hours-recurrences | 48 hours
  Time to the first documented AF recurrence excluding patients with recurrences in the first 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Vasilios Vasilikos, MD, Study Chair — 3rd University Cardiology Clinic of Ippokrateion Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart S, Hart CL, Hole DJ, McMurray JJ. Population prevalence, incidence, and predictors of atrial fibrillation in the Renfrew/Paisley study. Heart. 2001 Nov;86(5):516-21. doi: 10.1136/heart.86.5.516. PMID 11602543
- [Background] Aliot E, Capucci A, Crijns HJ, Goette A, Tamargo J. Twenty-five years in the making: flecainide is safe and effective for the management of atrial fibrillation. Europace. 2011 Feb;13(2):161-73. doi: 10.1093/europace/euq382. Epub 2010 Dec 7. PMID 21138930
- [Background] Anderson JL, Gilbert EM, Alpert BL, Henthorn RW, Waldo AL, Bhandari AK, Hawkinson RW, Pritchett EL. Prevention of symptomatic recurrences of paroxysmal atrial fibrillation in patients initially tolerating antiarrhythmic therapy. A multicenter, double-blind, crossover study of flecainide and placebo with transtelephonic monitoring. Flecainide Supraventricular Tachycardia Study Group. Circulation. 1989 Dec;80(6):1557-70. doi: 10.1161/01.cir.80.6.1557. PMID 2513143
- [Background] Naccarelli GV, Dorian P, Hohnloser SH, Coumel P. Prospective comparison of flecainide versus quinidine for the treatment of paroxysmal atrial fibrillation/flutter. The Flecainide Multicenter Atrial Fibrillation Study Group. Am J Cardiol. 1996 Jan 25;77(3):53A-59A. doi: 10.1016/s0002-9149(97)89118-7. PMID 8607392
- [Background] van Wijk LM, den Heijer P, Crijns HJ, van Gilst WH, Lie KI. Flecainide versus quinidine in the prevention of paroxysms of atrial fibrillation. J Cardiovasc Pharmacol. 1989 Jan;13(1):32-6. doi: 10.1097/00005344-198901000-00005. PMID 2468933
- [Background] Capucci A, Piangerelli L, Ricciotti J, Gabrielli D, Guerra F. Flecainide-metoprolol combination reduces atrial fibrillation clinical recurrences and improves tolerability at 1-year follow-up in persistent symptomatic atrial fibrillation. Europace. 2016 Nov;18(11):1698-1704. doi: 10.1093/europace/euv462. Epub 2016 Feb 17. PMID 26893497
- [Background] Fragakis N, Koskinas KC, Vassilikos V. Ranolazine as a promising treatment option for atrial fibrillation: electrophysiologic mechanisms, experimental evidence, and clinical implications. Pacing Clin Electrophysiol. 2014 Oct;37(10):1412-20. doi: 10.1111/pace.12486. Epub 2014 Aug 19. PMID 25138058
- [Background] Sicouri S, Glass A, Belardinelli L, Antzelevitch C. Antiarrhythmic effects of ranolazine in canine pulmonary vein sleeve preparations. Heart Rhythm. 2008 Jul;5(7):1019-26. doi: 10.1016/j.hrthm.2008.03.018. Epub 2008 Mar 21. PMID 18598958
- [Background] Burashnikov A, Di Diego JM, Zygmunt AC, Belardinelli L, Antzelevitch C. Atrium-selective sodium channel block as a strategy for suppression of atrial fibrillation: differences in sodium channel inactivation between atria and ventricles and the role of ranolazine. Circulation. 2007 Sep 25;116(13):1449-57. doi: 10.1161/CIRCULATIONAHA.107.704890. Epub 2007 Sep 4. PMID 17785620
- [Background] Murdock DK, Reiffel JA, Kaliebe J, Larrain G. The Conversion of Paroxysmal or Initial Onset Atrial Fibrillation with Oral Ranolazine: Implications for a New
- [Background] Fragakis N, Koskinas KC, Katritsis DG, Pagourelias ED, Zografos T, Geleris P. Comparison of effectiveness of ranolazine plus amiodarone versus amiodarone alone for conversion of recent-onset atrial fibrillation. Am J Cardiol. 2012 Sep 1;110(5):673-7. doi: 10.1016/j.amjcard.2012.04.044. Epub 2012 May 22. PMID 22621799
- [Background] Koskinas KC, Fragakis N, Katritsis D, Skeberis V, Vassilikos V. Ranolazine enhances the efficacy of amiodarone for conversion of recent-onset atrial fibrillation. Europace. 2014 Jul;16(7):973-9. doi: 10.1093/europace/eut407. Epub 2014 Jan 27. PMID 24473502
- [Background] De Ferrari GM, Maier LS, Mont L, Schwartz PJ, Simonis G, Leschke M, Gronda E, Boriani G, Darius H, Guillamon Toran L, Savelieva I, Dusi V, Marchionni N, Quintana Rendon M, Schumacher K, Tonini G, Melani L, Giannelli S, Alberto Maggi C, Camm AJ; RAFFAELLO Investigators (see Online Supplementary Appendix for List of Participating Centers and Investigators). Ranolazine in the treatment of atrial fibrillation: Results of the dose-ranging RAFFAELLO (Ranolazine in Atrial Fibrillation Following An ELectricaL CardiOversion) study. Heart Rhythm. 2015 May;12(5):872-8. doi: 10.1016/j.hrthm.2015.01.021. Epub 2015 Jan 17. PMID 25602175
- [Background] Kirstein M, Eickhorn R, Langenfeld H, Kochsiek K, Antoni H. Influence of beta-adrenergic stimulation on the fast sodium current in the intact rat papillary muscle. Basic Res Cardiol. 1991 Sep-Oct;86(5):441-8. doi: 10.1007/BF02190712. PMID 1662947
- [Background] Schubert B, Vandongen AM, Kirsch GE, Brown AM. Inhibition of cardiac Na+ currents by isoproterenol. Am J Physiol. 1990 Apr;258(4 Pt 2):H977-82. doi: 10.1152/ajpheart.1990.258.4.H977. PMID 2158748
- [Background] Burashnikov A, Sicouri S, Di Diego JM, Belardinelli L, Antzelevitch C. Synergistic effect of the combination of ranolazine and dronedarone to suppress atrial fibrillation. J Am Coll Cardiol. 2010 Oct 5;56(15):1216-24. doi: 10.1016/j.jacc.2010.08.600. PMID 20883928
- [Background] Sicouri S, Burashnikov A, Belardinelli L, Antzelevitch C. Synergistic electrophysiologic and antiarrhythmic effects of the combination of ranolazine and chronic amiodarone in canine atria. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):88-95. doi: 10.1161/CIRCEP.109.886275. Epub 2009 Dec 1. PMID 19952329